CLINICAL TRIAL: NCT03618914
Title: Interactive Effects of Iron Status and Inflammation on Serum Hepcidin and Erythrocyte Iron Incorporation in Young Women
Brief Title: Anemia and Inflammation
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Ibn Tofail University-CNESTEN (Unknown)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. Dr. med., Swiss Federal Institute of Technology
Other Study IDs: SMILE Study
Record Dates: First submitted 2018-07-23; First posted 2018-08-07 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Iron Deficiency Anemia; Inflammation
MeSH Terms: conditions — Anemia, Iron-Deficiency; Inflammation | interventions — vaxigrip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-anemic women
  Interventions: Biological: Dultavax and Vaxigrip
- anemic women: anemia due to iron deficiency
  Interventions: Biological: Dultavax and Vaxigrip

INTERVENTIONS:
Biological: Dultavax and Vaxigrip — All the women got an influenza/DTP vaccine in order to induce acute inflammation

SUMMARY:
During inflammation hepcidin concentrations are increased, leading to a decrease in iron absorption. In iron deficiency anemia hepcidin is suppressed due to the activation of erythropoiesis. Whether inflammation or anemia has the stronger effect on hepcidin is uncertain.

ELIGIBILITY:
Inclusion Criteria:

* BMI <27.5kg/m2
* body weight <70kg
* either non-anemic (Hb>12.5g/dl) or anemic (Hb between 8-12 g/dl and ferritin <15ng/ml)

Exclusion Criteria:

* pregnant or lactating
* chronic disease
* smoking
* inflammation defined as CRP<5mg/L; AGP<1g/L

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young women with or without iron-deficiency anemia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Fractional and total iron absorption | 14 days after the second baseline test meal administration
Fractional and total iron absorption | 14 days after the test meal administered 24 hours after vaccination

SECONDARY OUTCOMES:
Serum hepcidin | up to 36 hours
Serum Interleukin 6 | up to 36 hours
  inflammation
Serum ferritin | up to 36 hours
  Iron status
Serum transferrin | up to 36 hours
  Iron status
Serum CRP | up to 36 hours
  inflammation
Serum AGP | up to 36 hours
  inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Ibn Tofail University-CNESTEN, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: No